CLINICAL TRIAL: NCT04398225
Title: A Phase 1b, Multicenter, Open-label, Multiple Ascending Dose Trial to Assess the Pharmacokinetics, Safety and Tolerability of Centanafadine Extended-release Capsules After Oral Administration in Pediatric Subjects (4 to 12 Years, Inclusive) With Attention-deficit/Hyperactivity Disorder
Brief Title: A Trial to Assess the Pharmacokinetics, Safety, and Tolerability of Centanafadine in Pediatric Subjects With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00010
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (9-12 y) (Experimental): Centanafadine extended release capsule; 100 mg adult equivalent; twice daily for 14 days
  Interventions: Drug: Centanafadine
- Cohort 2 (9-12 y) (Experimental): Centanafadine extended release capsule; 200 mg adult equivalent; twice daily for 14 days
  Interventions: Drug: Centanafadine
- Cohort 3 (9-12 y) (Experimental): Centanafadine extended release capsule; 400 mg adult equivalent; twice daily for 14 days
  Interventions: Drug: Centanafadine
- Cohort 4 (6-8 y) (Experimental): Centanafadine extended release capsule; 100 mg adult equivalent; twice daily for 14 days
  Interventions: Drug: Centanafadine
- Cohort 5 (4-5 y) (Experimental): Centanafadine extended release capsule; 100 mg adult equivalent; twice daily for 14 days
  Interventions: Drug: Centanafadine

INTERVENTIONS:
Drug: Centanafadine — Extended release capsule

SUMMARY:
This trial will evaluate the pharmacokinetics, safety, and tolerability of centanafadine in pediatric subjects with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 4 to 12 years of age, inclusive, at the time of informed consent/assent.
* Subjects must weight ≥ 13 kg.
* Subjects with a diagnosis of any ADHD subtype based on Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria and confirmed by the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-Kid).
* Subject is judged by the investigator to be clinically stable, and has not had any psychiatric hospitalizations within the past 12 weeks.
* Subjects and their caregivers must be able and willing to utilize the AiCure Platform for each daily dose.

Exclusion Criteria:

* Subjects with a clinical presentation or history that is consistent with delirium, dementia, amnesia, or other cognitive disorders; subjects with psychiatric symptoms that are better accounted for by another psychiatric or general medical condition(s) or direct effect of a substance.
* Subjects with developmental disorders, such as Autism Spectrum Disorder.
* Subjects with a history of at least mild intellectual disability as determined by IQ < 70, clinical evidence, or a social or school history that is suggestive of intellectual disability.
* Subjects with hypothyroidism or hyperthyroidism (unless condition has been stabilized with medications for at least 90 days prior to first dose of IMP) or an abnormal result for free T4 at screening.
* Subjects who currently have clinically significant neurological, dermatological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV seropositive status/AIDS, or chronic hepatitis B or C.
* Subjects with insulin dependent diabetes mellitus (i.e. any subjects using insulin)
* Subjects with epilepsy, Tourette's Disorder, or a history of seizures or a history of severe head trauma or cerebrovascular disease.
* Any major surgery within 30 days prior to the first dose of IMP.
* Any history of significant bleeding or hemorrhagic tendencies.
* Blood transfusions within 30 days prior to the first dose of IMP.
* Subjects who have supine or standing diastolic blood pressure, after resting for at least 5 minutes, > 80 mmHg.
* Subjects who participated in a clinical trial and were exposed to IMP within the last 30 days prior to screening or who participated in more than 2 interventional clinical trials within the past year. Subjects who have had any previous exposure to centanafadine.
* Subjects with a history of true allergic response to a medication or a history of dermatologic adverse reactions or anaphylaxis secondary drug exposure.
* Subjects with a history of allergic reaction or known or suspected sensitivity to any substance that is contained in the IMP formulation.
* Subjects who do not tolerate venipuncture or have poor venous access that would cause difficulty for collecting blood samples.
* Consumption of alcohol and/or food and beverages containing methylxanthines, foods known to affect CYP1A2 (e.g. charbroiled or pan-fried meats and cruciferous vegetables) within 72 hours prior to dosing.
* Relative of the trial site employees cannot participate in the trial.
* Siblings, other family members, and those having the same place of residence as the subject are also excluded from the trial.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Maximal peak plasma concentration (Cmax) | 24 hours
Area under the concentration-time curve from time 0 to 24 hours (AUC0-24h) on day 14 | 24 hours
Apparent clearance and apparent volume of distribution of centanafadine on Day 14 | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com